CLINICAL TRIAL: NCT00516334
Title: Advanced Electrophysiological Studies of the Premature Newborn Infant Brain: Understanding Brain Injury
Brief Title: Study of Bedside EEG to Evaluate Brain Injury in Premature Newborns
Acronym: BrainZ
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Linda J. Van Marter, M.D., M.P.H., Attending Neonatologist and Associate Professor of Pediatrics Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: 2003-P-000088
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Brain Injury; Seizures; Cerebral Palsy
Keywords: brain; electroencephalography; premature infant; neurodevelopment
MeSH Terms: conditions — Brain Injuries; Seizures; Cerebral Palsy; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is evaluating whether a bedside brainwave monitor can be used to detect early brain injury in premature infants.

DETAILED DESCRIPTION:
Patient enrollment and electroencephalographic (EEG) and clinical data collection stopped May 2009. Data analysis is ongoing, and results have been described (O'Reilly D, Navakatikyan MA, Filip M, Greene D, Van Marter LJ. Peak to Peak Amplitude in Neonatal Brain Monitoring of Premature Infants. Clin Neurophysiol 2012 May 16), via publication in a peer-reviewed journal. Another manuscript has been completed and is undergoing revision for resubmission. We anticipate several additional articles will be completed from the data collected during this study. There is no relationship between industry and no current funding for this study. We maintain institutional review board approval due to ongoing data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Infants inborn below 28 weeks gestation

Exclusion Criteria:

* At birth, deemed not likely to survive 7 days or more
* Major intracranial congenital anomaly

Ages: 1 Day to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants <29 weeks gestational age
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Van Marter, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Deirdre O'Reilly, MD, MPH, Study Director — Boston Children's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States